CLINICAL TRIAL: NCT06126770
Title: Development and Testing of Balika Bodhu: a Social Norm Intervention to Address Denial of Sexual and Reproductive Health and Rights to Married Adolescent Girls in Rural Bangladesh
Brief Title: Development and Testing of Balika Bodhu
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Global Affairs Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-22145
Record Dates: First submitted 2023-10-12; First posted 2023-11-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Sexual and Reproductive Health and Rights
Keywords: Married adolescent girls; Sexual and reproductive health and rights; Family planning; Conception; SRH service uptake; Intimate Partner violence; Consent and choice; Critical consciousness; Empowerment; Agency; Social norms; Gender norm
MeSH Terms: conditions — Coitus; Empowerment

STUDY DESIGN:
Intervention Model Description: Mixed method 2-arm cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The social norm intervention (Experimental): The married adolescent girls (MAGs) and their spouses, and community members from the intervention clusters will receive the social norm intervention.
  Interventions: Behavioral: The social norm intervention
- Pure Control (No Intervention): Participants, including married adolescent girls (MAGs), their spouses, and community members from the control clusters, will not receive any intervention.

INTERVENTIONS:
Behavioral: The social norm intervention — The intervention will target Married adolescent girls, their spouses, and elderly/influential community members. Thirty-six 2-hour weekly sessions will be conducted with MAGs. The session topics will be categorized into two broad headings: i) Health and life skills sessions covering, for example topics such as sex and gender, rights, marriages, SRHR, and ii) Business and entrepreneurship sessions.
  Spouses of the MAGs will receive 20 2-hour bi-weekly sessions. A total of three 2-hour couples sessions will be held. Elderly women and influential community members will have three 2-hour bi-monthly sessions. In addition, MAGs with leadership qualities will be identified and trained to conduct campaigns and activism. They will also receive training on income generating.
  Arms: The social norm intervention

SUMMARY:
The study aims to generate knowledge on barriers experienced by married adolescent girls (MAGs) in demanding, accessing and practicing their rights regarding their sexual and reproductive health (SRH), including family planning (FP) use, conception, and seeking health care relating to SRH. We will also explore the underlying factors influencing such barriers. The study will develop and test a social norms intervention that addresses the gaps in programming and in the literature combining a comprehensive empowerment programme for MAGs with engagement of other stakeholders to increase demand, access and practices of positive behaviours in relation to sexual and reproductive health and rights (SRHR) among these girls. We will collaborate with a local organization, who usually work on empowerment and SRHR of women, for implementing the intervention and will build their capacity as well. The study will employ a mixed-method two-arm cluster randomized controlled trial design. All the information generated will inform the program and policy about the barriers and potential solutions to improve demand, access and practices of SRHR among the MAGs.

DETAILED DESCRIPTION:
Background Sexual and reproductive health and rights (SRHR) are vital to one's health and development. Over the last few decades Bangladesh, known as a patriarchal society, has made remarkable progress in improving contraceptive use, and maternal health. However, the progress has not been consistent in different SRHR domains and is not uniform across different groups of reproductive aged females. The progress was particularly slow in realising SRH rights of the women. Evidence suggests that choice and consent of females are ignored in all spheres of SRHR and that patriarchal gender and social norms, and discriminatory laws and practices in Bangladesh perpetuate denial of SRHR to females. Due to high prevalence of child marriage in Bangladesh (59%) (NIPORT & ICF, 2019) a huge proportion of adolescent girls are married before reaching 18. In a patriarchal setting such as Bangladesh with very strong gender and age hierarchies these child brides typically command the lowest power in the marital home. They typically have lower education than those who get married in adulthood. They also lack voice and bargaining skills. In such a context, the husband or mother-in-law may figure prominently in decisions about using contraception and the timing of childbearing. In this context, denial of SRHR usually becomes part of their lived experiences.

Although social norms are recognised as one of the main drivers of denial of SRHR to married adolescent girls (MAG), social norms theories and approaches to programming are relatively new and there has been little attempt to develop and rigorously test interventions to address such social norms worldwide and in Bangladesh. Also, a handful of programmes have been implemented worldwide and in Bangladesh to empower partnered female adolescents for promoting SRHR. But, we argue that conceptualization of empowerment in these initiatives were often not grounded in solid theory and evidence. Thus, empowerment programmes for women and girls often fail to include a critical component, namely, movement building and collective agency and critical consciousness, without which empowerment cannot take place in its true sense.

The current study proposes to develop and test Balika Bodhu, a social norm intervention to address the gaps in programming and in the literature combining a comprehensive empowerment programme for MAGs with engagement of other stakeholders to increase demand, access and practice of positive behaviours in relation to SRHR among these MAGs. Balika Bodhu covers married adolescent girls aged 15-19 years.

The Balika Bodhu intervention The Balika Bodhu intervention will be developed heavily drawing on CARE's IMAGINE model, and on SAFE, a project spearheaded by icddr,b and aimed at promoting SRHR and addressing violence against women in slums of Dhaka.

Balika Bodhu intervention will be implemented by Nari Maitree, an NGO working on women's issues. The research team will conduct both quantitative and qualitative monitoring for documenting implementation fidelity. Effectiveness of the intervention will be assessed in changing social norms endorsing denial of SRHR to MAGS and in empowering them to demand, access and practice SRHR. The intervention will involve a 12-month gender transformative participatory programming for: (1) empowering MAGs and (2) creating an enabling environment in the family and the community for the MAGs to demand, access and practice SRHR.

The intervention will target Married adolescent girls, their spouses, and elderly/influential community members. Thirty-six 2-hour weekly sessions will be conducted with MAGs. The session topics will be categorized into two broad headings: i) Health and life skills sessions covering, for example topics such as sex and gender, rights, marriages, SRHR (e.g., first conception, birth spacing, contraception, healthy relationships, polygamy, divorce, gender-based violence (GBV), communication and negotiation, anger and conflict management, goal setting, household budgeting, activism, leadership skills, and community action planning, and ii) Business and entrepreneurship sessions, which will basically include sessions smart planning of businesses (e.g., market research, business planning, and adding value).

Spouses of the MAGs will receive 20 2-hour bi-weekly sessions. The session topics will cover: sex and gender, rights, marriages, registration, dowry, conception and contraception, healthy relationships, polygamy, divorce, gender-based violence (GBV), communication and negotiation, anger and conflict management, goal setting, and household budgeting.

A total of three 2-hour couples sessions will be held, each to be delivered every two months, starting from the 6th month of the intervention. The session topics will include teenage pregnancy, unwanted pregnancy, and action planning. Elderly and influential community members will have three 2-hour bi-monthly sessions starting from the 6th month of the intervention, covering topics related to teenage pregnancy, unwanted pregnancy, and action planning.

MAGs with leadership qualities will be identified and trained to conduct campaigns and activism. They will be put in contact with other girls' groups and networks, mentored and given access to resources to execute four community-level social norm activities. These leaders will also receive training on income generating.

Hypothesis Balika Bodhu, a social norm intervention on sexual and reproductive health and rights (SRHR) combining a comprehensive empowerment package for married adolescent girls (MAGs) and positive engagement of relevant stakeholders will significantly improve demand, access and practices regarding SRHR among MAGs in family planning (FP) use, conception, and SRH service uptake.

Objectives

Primary objective:

1. To develop Balika Bodhu, a social norm intervention combining empowerment of MAGs and mobilisation of relevant stakeholders to promote demand for, access to, and practices of SRHR, including FP use, conception and SRH service uptake.
2. To measure the effect of Balika Bodhu in increasing demand for, access to, and practices of SRHR (FP use, conception, and SRH service uptake) of MAGS.

   Secondary objectives:
3. To measure the effect of Balika Bodhu on empowerment of MAGs;
4. To measure the effect of Balika Bodhu on social norm regarding SRHR of MAGs;
5. To explore how change happens or why change does not occur.

Methods Study design Balika Bodhu will involve a mixed-method two-arm (intervention and control) Cluster Randomized Controlled Trial (CRCT) design.

Study site Balika Bodhu will be implemented in 32 clusters (villages, primary sampling unit) in Rajbari Sadar upazila of Rajbari district.

Cluster formation and randomization The villages from Rajbari Sadar upazila will be treated as clusters or the primary sampling units in this study. Thirty-two clusters will be formed ensuring sufficient buffer zone around each cluster, and then will be randomized to two study arms (intervention and control).

Household enumeration, sampling, recruitment of study participants and survey and qualitative data collection Once the clusters have been selected and randomized to intervention and control arms, an enumeration of the households in each cluster will be conducted to collect socio-demographic information on the household members (e.g., sex, date of birth, age and marital status) to form the sampling frame for the MAGs', their husbands' and the community survey.

A total of 1120 MAGs will be randomly selected (35 per cluster) from the list obtained through household enumeration. Their husbands will also be included in the study. Upon receiving consent, the selected MAGs and their husbands will be enrolled in the study and included in the baseline survey. Following the baseline survey interviews, MAGs from the intervention villages will be invited to participate in the Balika Bodhu intervention, and upon receiving their consent, they will be formally enrolled in the intervention. All MAGs and their husbands who were interviewed at baseline will also be targeted for follow-up interviews at the endline.

For the community survey, separate cross-sectional samples will be drawn and interviewed at baseline and endline. We will obtain lists of eligible community members (females and males), aged 35 years or more from household enumeration. Nine females and nine males will be randomly selected from each cluster for inclusion in the surveys making the total in each round 576.

Qualitative data will be collected at baseline and endline from two intervention clusters using 32 In-depth Interviews (with 16 MAGs and 16 husbands of MAGs), and 6 Key Informant Interviews (with mothers-in-law of MAGs, NGO staff, CHWs, village doctors/ traditional healers/ drug sellers) and 8 Focus Group Discussions (with MAGs, their spouses, and elderly women/influential community members aged 35 years or more).

Blinding No one will be blinded during this selection and allocation process in this study.

Quantitative data analyses During baseline we will explore the current situation in empowerment and SRHR among MAGs and their correlates, while at end line we will measure the impact of the social norms intervention on empowerment, on social norm change and promotion of demand, access and positive practices in relation to SRHR among the MAGs. Descriptive analyses will be performed to report frequencies and percentages of different outcomes of interest. Chi-square, ANOVA and t-tests will be performed to check whether the study arms are covariate balanced. Linear and logistic regression analyses will be performed to identify the underlying factors for current situation in SRHR among MAGs.

Intention-to-treat (ITT) analysis will be used during assessing the impact of the intervention. Thus, all the MAGs enrolled at baseline and could be successfully interviewed at endline will be included in the analysis irrespective of their actual level of participation in the intervention activities. The information on participation of study participants in the intervention activities will come from the programme monitoring data and will also used in the models. The impact of the intervention on primary and secondary outcomes will be assed using risk ratios/regression coefficients derived from binary/linear regression analyses for measuring change in outcomes in the intervention arms relative to change in the control arm. Significance level will be set at p<.05 for all analyses. The data will be analysed using STATA 16.

Qualitative data analyses With the informants' permission, all interviews and FGDs will be digitally recorded. All recorded interviews will be transcribed verbatim. Data analysis will be iterative. To explore research questions, we will combine the intense, within-case focus of Narrative Analysis with the across-case approach of Grounded Theory, a robust analytic strategy for qualitative data.

Ethical considerations This study will be guided by CIOMS International Guidelines for Ethical Review of Epidemiological Studies and the WHO recommendations for ethical considerations in researching violence against. The study will seek ethical approval from icddr,b's institutional review board. This application and all documents related to the protection of human subjects will be reviewed the IRB of icddr,b. All members of the research team will be trained to meet the highest ethical standards of data collection and analysis.

The MAGs who are minor (aged below 18) will be considered as "mature minors" and informed consent will be sought by the interviewer prior to the interview with each study participant. Participation in the study will be as entirely voluntary. All the participants will be informed orally of the purpose and nature of the study, its expected benefits, sensitivity, confidentiality and voluntary nature of participation.

ELIGIBILITY:
Inclusion criteria:

For MAGs:

i) Adolescent girls aged 15-19 years; ii) Currently married and living with husband; and iii) Both the girl and her husband have no intention of migrating out within the next 15 months.

For husbands:

i) The husbands of the selected adolescent girls will also be eligible to be included in the study.

For community members:

i) Aged 35-59 years.

Exclusion criteria:

i) MAGs who are physically or mentally unstable; ii) Any couple having plans to migrate out during the next one and a half years.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2918 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Instrumental agency of MAGs in decision making regarding SRHR | 15 months
  The MAGs will be asked about who was the main decision maker regarding: (a) FP use; (b) timing of first conception; and (c) number of children to have. The response options included "1=the MAG herself", "2=husband", "3=jointly" and "4=someone else". A follow up question, "what kind of joint decision it was", was asked in every case when the respose was "jointly". The response options included "1=he said about his choice and I agreed", "he said his choice and forced me to agree", and "3=I said my choice and he agreed". A MAG will be considered having the agency in decision making regarding a specific theme of SRHR and will be coded as "Yes=1" if she decided herself or it was a joint decision without any force on her, and "No=2" otherwise. We will generate a summative score, with higher score indicating higher agency. The score will then be divided into tertiles.

SECONDARY OUTCOMES:
Intrinsic agency of MAGs | 15 months
  We will assess women's intrinsic agency, using a validated, 29-item three-dimensional measure capturing women's intrinsic voice and mobility; gender equitable attitudes; and non-justification of wife beating (CFA standardized factor loadings: 0.54-0.81, 0.35-0.82, and 0.87-0.93, respectively; CFI = 0.94; TLI = 0.93; RMSEA = 0.04). Summative scores will be obtained. Negatively valenced items will be reverse-coded, so higher scores indicates higher agency.
Instrumental agency of MAGs | 15 months
  We will assess women's instrumental agency using a validated, 17-item three-dimensional measure capturing women's use of financial services, voice with husband, and voice and mobility outside the home (CFA standardized loadings 0.57-0.95, 0.48-0.99, and 0.43-0.79, respectively, CFI = 0.94, TLI = 0.93, RMSEA = 0.05). Summative scores will be obtained. Negatively valenced items will be reverse-coded, so higher scores indicates higher agency.
Collective agency of MAGs | 15 months
  We will assess women's collective agency regarding influence in the community using an eight-item validated scale (CFA standardized loadings 0.52-0.84; CFI = 0.96; TLI = 0.95; RMSEA = 0.10) and regarding women's leadership in groups using a validated seven-item scale (CFA standardized loadings: 0.54-0.83; CFI = 0.96; TLI = 0.95; RMSEA = 0.10). The participants will report their agreement (1 = totally disagree to 4 = totally agree) with statements like "women like me can really understand what is going on with my community" and "I am often a leader in groups," "I prefer to be a leader rather than a follower," and "Other people usually follow my ideas", etc. Summative scores will be obtained. Negatively valenced items will be reverse-coded, so higher scores indicates higher collective agency.
Critical Consciousness of MAGs related to their consent and choice in SRH | 15 months
  Critical Consciousness is theorized to be composed of two subcomponents. The critical reflection component encompasses critically reflecting on perceived societal inequalities as well as the endorsement of societal equality; the critical action component encompasses individual or collective action taken to change perceived social inequalities. We will measure the critical consciousness of MGAs using the validated 15-item Critical Consciousness Scale. Ten critical reflection related items will be used to measure the perceived inequality and egalitarianism. The response options include: strongly agree, agree, disagree and strongly disagree. Another five items will be used to assess critical action, or the degree to which they have participated in individual and/or collective action to produce socio political change, with the response options - not at all, rarely, sometimes and often. A summative score will be obtained, with higher score indicating higher critical consciousness.
Knowledge of MAGs regarding SRHR | 15 months
  The MAGs will be asked two questions about their knowledge regarding FP: i) which of the FP methods have you heard of?; and ii) have you heard about emergency contraceptive pill?. Their knowledge will be measured in terms of their report on number of modern methods, and emergency contraceptive pill.
  The MAGs will be asked four questions about their knowledge regarding conception. Their knowledge will be measured in terms of their report of correct knowledge on: i) appropriate age at first conception for a woman; and ii) possibility of a woman becoming pregnant before her menstrual period has returned after the birth of a child; iii) number of potential problems regarding teenage pregnancy; and iv) number of consequences in case of not having proper spacing between two pregnnacies.
Positive attitudes of MAGs regarding SRHR | 15 months
  Attitudes of MAGs regarding SRHR will be measured using six items, like "family planning is a women's business and a man should not worry" and "a woman has right to choose when to first conceive". The participants will report their agreement on a likert scale (1 = strongly agree to 4 = strongly disagree). A summative score will be obtained, with higher score indicating more positive attitude regarding SRHR. The score will then be divided into tertiles.
Couple communication initiated by MAGs regarding their SRHR | 15 months
  The MAGs will be asked whether she had any communication/discussion with her husband regarding FP use, first conception, and number of children they want to have. The response options include "1=Yes" and "2=No". They will also be asked about who started the conversation, with the response options "1=herself", "2=husband" and "3=don't remember". A MAG will be considered initiated the couple communication if there was a conversation which was started by the MAG herself regarding any specific SRHR issue, and will be coded as "Yes=1", and "No=0" otherwise. A summative score will be obtained by accumulating the number of conversations she initiated on different SRHR issues, with higher score indicating higher partner commnunication. The score will then be divided into tertiles.
MAGs attempts to negotiate their choice regarding SRHR | 15 months
  The MAGs will be asked about what happened if there was any mismatch between her and her husband's choice regarding the above mentioned SRHR themes. For instances, i) what was her reaction; ii) what was her husband's reaction; iii) whether she accepted her husband's choice or her husband accepted her choice, etc. A MAG will be considered having an attempt to negotiate if she tried to negotiate her choice with her husband regarding any specific SRHR issue, and will be coded as "Yes=1", and "No=0" otherwise. A summative score will be obtained by accumulating the number of SRHR themes where she could acheive her own choice, with higher score indicating better negotiation skill. The score will then be divided into tertiles.
SRH service uptake among MAGs | 15 months
  If any MAG reports having an induced abortion/MR, she will asked about place, provider and the method of abortion. The MAGs will be asked about the post-abortion care irrespective of whether it was an induced or spontaneous abortion. The MAGs who report experiencing any physical and/or sexual intimate partner violence will be asked about help seeking. The results will be presented in frequencies and percentages.
Prevalence of intimate partner violence among MAGs | 15 months
  MAGs' experience of IPV (i.e. controlling behaviour, and physical and sexual violence IPV) will be measured using a modified version of The Revised Conflict Tactic Scale. The scale is the most widely used measure of IPV which is characterized by having direct and behaviourally explicit questions in order to reduce variation in the interpretation and understanding of what violence comprises of. These instruments are designed to minimize reporting biases that arise from subjective perceptions of abuse by asking only about specific behaviours perpetrated by a male partner. To measure economic coercion, we will use a modified version of the ECS-20.. A woman will be considered exposed to any specific type of IPV if she responds "yes" to any of the items related to that specific type of IPV, and will be coded "yes=1", and "no=0" otherwise.
Knowledge of husbands of MAGs regarding SRHR of MAGs | 15 months
  The husbands of MAGs will be asked two questions about their knowledge regarding FP: i) which of the FP methods have you heard of?; and ii) have you heard about emergency contraceptive pill?. Their knowledge will be measured in terms of their report on number of modern methods, and emergency contraceptive pill.
  The husbands of MAGs will be asked four questions about their knowledge regarding conception. Their knowledge will be measured in terms of their report of correct knowledge on: i) appropriate age at first conception for a woman; and ii) possibility of a woman becoming pregnant before her menstrual period has returned after the birth of a child; iii) number of potential problems regarding teenage pregnancy; and iv) number of consequences in case of not having proper spacing between two pregnancies.
Positive attitudes of husbands of MAGs regarding SRHR | 15 months
  Attitudes of husbands of MAGs regarding SRHR will be measured using six items, like "family planning is a women's business and a man should not worry" and "a woman has right to choose when to first conceive". The participants will report their agreement on a likert scale (1 = strongly agree to 4 = strongly disagree). A summative score will be obtained, with higher score indicating more positive attitude regarding SRHR. The score will then be divided into tertiles.
Positive attitudes regarding agency of MAGs regarding SRHR among their husbands | 15 months
  Attitudes of husbands of MAGs about agency of MAGs regarding SRHR will be measured using 12 items. A typical example includes "It should be a wife's decision when to have a child". The participants will report their agreement on a 4-point likert scale (1 = strongly agree to 4 = strongly disagree). A summative score will be obtained, divided into tertiles. Negatively valenced items will be reverse-coded, so higher score indicates more positive attitudes.
Positive attitudes of husbands of MAGs regarding violence against women | 15 months
  Attitudes of husbands of MAGs regarding violence against women will be measured using six items. A typical example includes "There are times when a woman deserves to be beaten". The participants will report their agreement on a 4-point likert scale (1 = strongly agree to 4 = strongly disagree). A summative score will be obtained, with higher score indicating more positive attitudes. The score will then be divided into tertiles.
Positive attitudes of husbands of MAGs regarding gender roles within household | 15 months
  Attitudes of husbands of MAGs regarding gender roles within household will be measured using three items. A typical example includes "Child care activies such as cleaning after toilet, giving bath is a mother's responsibility". The participants will report their agreement on a 4-point likert scale (1 = strongly agree to 4 = strongly disagree). A summative score will be obtained, with higher score indicating more positive attitudes. The score will then be divided into tertiles.
Knowledge of community member regarding SRHR of MAGs | 15 months
  The community members will be asked two questions about their knowledge regarding FP: i) which of the FP methods have you heard of?; and ii) have you heard about emergency contraceptive pill?. Their knowledge will be measured in terms of their report on number of modern methods, and emergency contraceptive pill.
  The community members will be asked four questions about their knowledge regarding conception. Their knowledge will be measured in terms of their report of correct knowledge on: i) appropriate age at first conception for a woman; and ii) possibility of a woman becoming pregnant before her menstrual period has returned after the birth of a child; iii) number of potential problems regarding teenage pregnancy; and iv) number of consequences in case of not having proper spacing between two pregnancies.
Positive attitudes of community members regarding SRHR | 15 months
  Attitudes of community members regarding SRHR (FP and conception) will be measured using six items, like "family planning is a women's business and a man should not worry" and "a woman has right to choose when to first conceive". The participants will report their agreement on a likert scale (1 = strongly agree to 4 = strongly disagree). A summative score will be obtained, with higher score indicating more positive attitude regarding SRHR. The score will then be divided into tertiles.
Positive attitudes of community members regarding agency of MAGs regarding SRHR | 15 months
  Attitudes of community members about agency of MAGs regarding SRHR will be measured using 12 items. A typical example includes "It should be a wife's decision when to have a child". The participants will report their agreement on a 4-point likert scale (1 = strongly agree to 4 = strongly disagree). A summative score will be obtained, divided into tertiles. Negatively valenced items will be reverse-coded, so higher score indicating more positive attitudes.
Positive attitudes of community members regarding violence against women | 15 months
  Attitudes of community members regarding violence against women will be measured using six items. A typical example includes "There are times when a woman deserves to be beaten". The participants will report their agreement on a 4-point likert scale (1 = strongly agree to 4 = strongly disagree). A summative score will be obtained, with higher score indicating more positive attitudes. The score will then be divided into tertiles.
Positive attitudes of community members regarding gender roles within household | 15 months
  Attitudes of community members regarding gender roles within household will be measured using three items. A typical example includes "Child care activies such as cleaning after toilet, giving bath is a mother's responsibility". The participants will report their agreement on a 4-point likert scale (1 = strongly agree to 4 = strongly disagree). A summative score will be obtained, with higher score indicating more positive attitudes. The score will then be divided into tertiles.
Community social norms regarding SRHR of MAGs | 15 months
  Social norms will be explored both among the MAGs and the community members around SRHR of MAGs (i.e., FP, conception, number of children, abortion and SRH service seeking). A set of questions will be formulated about empirical and normative expectations and will be used as a scale. The participants will report their agreement on a Likert scale (1 = totally disagree to 4 = totally agree). The scale will be validated using factor analysis before use. Once the final scale is constructed, a summative score will be obtained, with higher score indicating stronger positive social norm. The score will then be divided into tertiles.

CONTACTS AND LOCATIONS:
Overall Officials: Ruchira Tabassum naved, PhD, Principal Investigator — Emeritus Scientist
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Mamun MA, Mahmud S, Antu JF, Talukder A, Naved RT. A protocol for a cluster randomized controlled trial to assess the impact of Balika Bodhu: A combined empowerment and social norm based sexual and reproductive health and rights intervention for married adolescent girls in rural Bangladesh. PLoS One. 2024 Aug 23;19(8):e0304988. doi: 10.1371/journal.pone.0304988. eCollection 2024. PMID 39178272